CLINICAL TRIAL: NCT05706974
Title: Prospective Evaluation of Clinical Study Experiences of Patients With Bile Duct Cancer
Brief Title: Looking At Bile Duct Cancer Patient Experience Patterns in Medical Trials
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 81185723
Record Dates: First submitted 2023-01-20; First posted 2023-01-31 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-01

CONDITIONS: Bile Duct Cancer
Keywords: bile duct; bile duct cancer
MeSH Terms: conditions — Bile Duct Neoplasms

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Clinical trials can sometimes favor certain demographic groups. Additionally, there is limited research that delves into the factors that influence participation in clinical trials, both positive and negative.

The goal is to identify the obstacles and challenges that prevent participation in bile duct cancer clinical trials, as well as the reasons for withdrawal or discontinuation.

The insights gained from this study will ultimately benefit those with bile duct cancer who may be invited to participate in medical research in the years to come.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Signed written informed consent
* Patient has been diagnosed with bile duct cancer

Exclusion Criteria:

* Woman pregnant or susceptible to the being
* Inability to perform regular electronic reporting
* Inclusion in another investigational clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Bile duct cancer patients who are actively considering participating in an observational medical study, but have not yet completed enrollment and randomization.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Number of bile duct cancer patients who decide to enroll in a clinical study | 3 months
Rate of bile duct cancer patients who remain in a clinical study to completion | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Norton RA, Foster EA. Bile duct cancer. CA Cancer J Clin. 1990 Jul-Aug;40(4):225-33. doi: 10.3322/canjclin.40.4.225. PMID 2114201
- [Background] Ebata T, Hirano S, Konishi M, Uesaka K, Tsuchiya Y, Ohtsuka M, Kaneoka Y, Yamamoto M, Ambo Y, Shimizu Y, Ozawa F, Fukutomi A, Ando M, Nimura Y, Nagino M; Bile Duct Cancer Adjuvant Trial (BCAT) Study Group. Randomized clinical trial of adjuvant gemcitabine chemotherapy versus observation in resected bile duct cancer. Br J Surg. 2018 Feb;105(3):192-202. doi: 10.1002/bjs.10776. PMID 29405274
- [Background] Xiang YJ, Sun JX, Wu JY, Wang K, Feng JK, Wei YG, Zhou JY, Zhang ZB, Zhang YQ, Qin YY, Yan ML, Cheng SQ. Recurrence hazard rate in patients with hepatocellular carcinoma and bile duct tumor thrombus: a multicenter observational study. HPB (Oxford). 2022 Oct;24(10):1703-1710. doi: 10.1016/j.hpb.2022.04.007. Epub 2022 Apr 22. PMID 35523655

DOCUMENTS (1):
  • Informed Consent Form (2023-01-20): https://cdn.clinicaltrials.gov/large-docs/74/NCT05706974/ICF_000.pdf